CLINICAL TRIAL: NCT01460641
Title: Perfusion CT as a Predictor of Treatment Response in Patients With Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Aya Kamaya, Associate Professor of Radiology, Stanford University
Other Study IDs: REC0006; SU-10202011-8538 (Other: Stanford University); 19224 (Other: Stanford IRB)
Record Dates: First submitted 2011-10-21; First posted 2011-10-27 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — If the patient undergoes surgery to remove the lesion in the rectum, the surgical specimen will be examined by the pathologist, who will perform a variety of tests to detect evidence of new blood vessel growth. The sample will be stored per routine protocol of the Stanford Department of Pathology.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CT perfusion

SUMMARY:
A research study of rectal cancer perfusion (how blood flows to the rectum over time). We hope to learn whether perfusion characteristics of rectal masses may be predictive of response to treatment and whether rectal perfusion characteristics can be used to follow response to treatment.

DETAILED DESCRIPTION:
Recent advances in computed tomography (CT) technology have made CT perfusion imaging feasible for the assessment of tumor perfusion in solid tumors of the abdomen. CT perfusion has shown promising results in serving as a noninvasive method of predicting response to therapy in cancer patients. CT perfusion parameters have also been found to correlate with immunohistologic markers of angiogenesis in a number of solid tumors, suggesting a possible role for CT perfusion as a noninvasive biomarker of tumor angiogenesis. The goals of the investigators study are twofold: first, to determine the relationship between baseline CT perfusion characteristics of rectal cancers and their response to treatment, and second, to determine if perfusion CT can be used to subsequently monitor tumor response to treatment. The investigators hope to enroll those patients with locally advanced rectal cancer undergoing standard CT for pre-treatment planning, integrating CT perfusion imaging into the current abdomen/pelvis imaging protocol with close clinical and radiologic follow-up after treatment to determine response to therapy and time to disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or biopsy-proven, locally advanced rectal cancer will be eligible for enrollment.
* Patients must be 18 years or older. Patients must not be pregnant and, if of child-bearing age, must take precautions not to become pregnant.
* No life expectancy restrictions.
* ECOG and Karnofsky Performance Status will not be employed.
* Patients with renal failure are ineligible for this study (GFR must be > 60)
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have undergone prior treatment for rectal cancer are ineligible for enrollment.
* No restrictions regarding use of other investigational agents.
* Patients with severe contrast allergy are ineligible.
* Patients who are pregnant or are trying to become pregnant are excluded from this study.
* Patients who are cancer survivors or HIV-positive will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer undergoing standard CT for pre-treatment planning
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2016-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Tumor stage change from Computed Tomography (CT) perfusion measurement | 3 months

SECONDARY OUTCOMES:
Tumor perfusion as measured by perfusion CT. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States